CLINICAL TRIAL: NCT03348696
Title: A Multi-Centre Randomised Study Comparing Tapering Low Dose Dexamethasone to Other Standard of Care Therapies for Taxane- Associated Pain Syndrome (TAPS) in Breast Cancer Patients (OTT 17-02 REaCT-TAPS)
Brief Title: Comparing Tapering Low Dose Dexamethasone to Other Standard of Care Therapies for TAPS in Breast Cancer Patients
Acronym: REaCT-TAPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OTT 17-02
Record Dates: First submitted 2017-09-27; First posted 2017-11-21 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Early-stage Breast Cancer; Pain Syndrome
MeSH Terms: conditions — Breast Neoplasms; Somatoform Disorders | interventions — dexamethasone 21-phosphate; dexamethasone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dexamethasone tapering dose (Active Comparator): standard dexamethasone pre-medication (8mg B.I.D x 3 days commencing the day before chemotherapy) then 4mg 1x/d for 2 days followed by 2mg 1x/d for 2 days
  Interventions: Drug: Dexamethasone tapering dose
- dexamethasone physician choice (Active Comparator): standard dexamethasone pre-medication (i.e. 8mg B.I.D x 3 days commencing the day before chemotherapy) then physician choice interventions
  Interventions: Drug: Dexamethasone physician choice

INTERVENTIONS:
Drug: Dexamethasone tapering dose — dexamethasone standard of care pre-medication + dexamethasone tapering dose
  Other Names: dexamethasone sodium phosphate; dexamethasone acetate
  Arms: dexamethasone tapering dose
Drug: Dexamethasone physician choice — Dexamethasone standard of care pre-medication + dexamethasone physician choice
  Other Names: dexamethasone sodium phosphate; dexamethasone acetate
  Arms: dexamethasone physician choice

SUMMARY:
The REaCT TAPS clinical trial will compare a tapering dose of dexamethasone to other standards of care on the presence of taxane-associated pain syndrome (TAPS) in early stage breast cancer.

DETAILED DESCRIPTION:
Taxanes such as docetaxel and paclitaxel are widely used chemotherapeutic agents in patients with early stage breast cancer and is commonly associated with taxane-associated pain syndrome (TAPS). TAPS is characterized by disabling pain which usually starts a few days after taxane administration and lasting 2-5 days, often returning following subsequent chemotherapy treatments. TAPS can significantly reduce a patients quality of life, lead to requirements for potent analgesics, as well as dose reductions/delays or discontinuation of chemotherapy. There is currently no clinical guidelines for the optimal standard of care for the management and prevention of TAPS. This REaCT clinical trial investigates the optimal management of TAPS with a tapering dose of dexamethasone (standard premedication comprising 8mg twice daily for 3 days followed by 4mg once a day for 2 days followed by 2mg once a day for 2 days) compared to other standard of care management (i.e. standard premedication with 8mg dexamethasone twice daily for 3 days) as directed by the treating physician. This study will use an "integrated consent model" that involves "oral consent" rather than a written informed consent writing process.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving docetaxel-based chemotherapy (Docetaxel 75mg/m2 and cyclophosphamide once every 21 days; or Docetaxel 75mg/m2 and carboplatin and trastuzumab once every 21 days or Fluoro-uracil, epirubicin and cyclophosphamide for 3 cycles once every 21 days, then docetaxel 100mg/m2 once every 21 days; or Adriamycin and cyclophosphamide for 3 cycles, then docetaxel 100mg/m2 once every 21 days) for early stage breast cancer.

  * English literacy and ability to complete questionnaire
  * ≥19 years of age

Exclusion Criteria:

* Contraindication to dexamethasone
* Unable to give informed consent
* Prior receipt of taxane-based chemotherapy
* Patient has a significant emotional or psychiatric disorder that in the opinion of the investigator precludes study entry.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of TAPS | Change in TAPS from Days 1-7, 3 weeks
  TAPS will be evaluated using the validated Functional Assessment of Cancer Therapy (FACT)-Taxane questionnaire which rates physical, social/family, emotional and functional well being on a scale of 0 (not at all) to 4 (very much)

SECONDARY OUTCOMES:
Quality of Life | Time Frame: Days 1,3,5,7 and 3 weeks
  Quality of Life will be evaluated using the FACT-Taxane questionnaire which rates physical, social/family, emotional and functional well being on a scale of 0 (not at all) to 4 (very much)
Quality of Life | Time Frame: Days 1,3,5,7 and 3 weeks
  Quality of Life will be evaluated using the Memorial Symptom Assessment Scale (MSAS) which measures prevalence (scale 1 (rarely) to 4 (almost constantly), severity (scale 1(slight) to 4 (very severe)) and level of distress (scale 0 (none) to 4 (very much)) of symptoms on a scale of 1-4
Pain scores | Time Frame: Days 1,3,5,7 and 3 weeks
  Pain scores will be evaluated using the Brief Pain Inventory (BPI), which assesses the severity of pain on a scale of 1 (no pain) to 10 (worst pain imaginable), and relief of pain treatments on a scale of 0% (no relief) to 100% (complete relief)
Use of rescue analgesic | Time Frame: Days 1,3,5,7, 3 weeks
  requirement of use of rescue analgesics will be assessed by daily morphine equivalent dosing
Symptoms and signs associated with dexamethasone | baseline and Day 7
  this will be evaluated using the dexamethasone questions of the FACT-T questionnaire which asks questions specific to symptoms associated with dexamethasone on a scale of 0 (not at all) to 4 (very much)
Cost effectiveness | baseline and Day 7
  Incremental cost, incremental quality-adjusted life years (QALYs) and incremental cost effectiveness will be be evaluated using the EuroQol (EQ)-5D-5L questionnaire. This scale evaluates quality of life (mobility, self-care, pain/discomfort, anxiety) on a scale of 1 (no problem)-5 (severe problem)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Clemons, MD, Principal Investigator — Ottawa Hospital Cancer Centre
Locations (2):
- Canada (2):
  - Southlake Regional Cancer Centre, Newmarket, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clemons M, Simos D, Sienkiewicz M, Ng T, Zibdawi L, Basulaiman B, Awan A, Fergusson D, Vandermeer L, Saunders D, Hutton B, Amir E; REThinking Clinical Trials (REaCT) Investigators. A prospective multi-centre, randomized study comparing the addition of tapering dexamethasone to other standard of care therapies for taxane-associated pain syndrome (TAPS) in breast cancer patients. Support Care Cancer. 2021 Oct;29(10):5787-5795. doi: 10.1007/s00520-021-06142-8. Epub 2021 Mar 19. PMID 33742240